CLINICAL TRIAL: NCT01932671
Title: Optimising Risk Assessment With CT-angiography or Calcium Score in Patients at High Risk for a Cardiovascular Event
Brief Title: The SMART-ORACLE Study
Acronym: SMART-ORACLE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. dr. Y. van der Graaf, Prof. dr. Y. van der Graaf, UMC Utrecht
Other Study IDs: NL36828.041.11
Record Dates: First submitted 2013-08-18; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease; Stroke; Peripheral Arterial Disease; Hypertension; Diabetes Mellitus, Type 2
Keywords: Cardiovascular diseases; Atherosclerosis; Multidetector Computed Tomography; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Coronary Artery Disease; Stroke; Peripheral Arterial Disease; Hypertension; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SMART: The SMART (Second Manifestation of ARTerial disease) cohort comprises patients at high-risk for or who have clinically manifest cardiovascular disease, including transient ischemic attack, cerebrovascular disease, peripheral artery disease, aneurysma aorta abdominalis, myocardial infarction, coronary ischemia for which coronary intervention is required, renal artery stenosis, diabetes mellitus, hyperlipidemia, hypertension, patients diagnosed with human immunodeficiency virus, pre-eclampsia, HELLP syndrome, abruption placentae and Intrauterine growth restriction in medical history. Participants are re-invited after 4 years for a second screening. This screening is performed to study the progression of atherosclerosis and evaluate the effects of the advice of the multidisciplinary team.

SUMMARY:
After having had a first cardiovascular event, there is a considerable risk of developing a subsequent event. Only recently, a risk prediction model was developed for this group of patients. Imaging techniques such as the coronary artery calcium score and contrast-enhanced computed tomography (CT) of the coronary and carotid arteries could be able to add improve this model. Imaging may further improve the prediction of future manifestations of arterial disease and personalize disease monitoring and treatment.

DETAILED DESCRIPTION:
Patients with a prior cardiovascular event exhibit an elevated risk for subsequent cardiovascular events. The Second Manifestation of Arterial Disease Study (SMART) has recruited over 10,000 patients since 1996 with clinically manifest cardiovascular disease in a multidisciplinary single center study involving primary care physicians, cardiologists, neurologists, vascular surgeons, vascular medicine specialists and radiologists. Within this study a prediction model was developed to accurately estimate the risk for new cardiovascular events. It is now possible to acquire high-quality motion-free computed tomography (CT) images of the coronary and carotid arteries. Imaging biomarkers extracted from these images may further improve the prediction of future manifestations of arterial disease and personalize disease monitoring and medical care.

The SMART-ORACLE study is a prospective, single center, observational cohort study aiming to include 1500 patients. The primary aim is to identify predictors of future cardiovascular events. Eligible patients will be selected via the recruitment of the original SMART study. Patients participating in the SMART-ORACLE study will undergo calcium scoring in multiple cardiovascular beds and contrast-enhanced CT-scans of the coronary and carotid arteries in addition to the regular SMART investigations. Patients with renal dysfunction will be either excluded from the study or will receive pre-hydration (depending on eGFR) to minimize the risk of contrast nephropathy. Follow-up with questionnaire-based assessment will take place every 26 weeks until death of participant or end of the SMART study, asking participants about possible new cardiovascular events. Endpoints will be adjudicated by a committee of three experts. The aim is to collect 170 future events.

The main analysis will consist of Cox proportional hazard analysis. Imaging biomarkers will be added to the existing prediction model to assess their (independent) discriminatory capacity for future events. The c-statistic will be used to measure the discrimination of each model. Net reclassification improvement tables will be constructed to evaluate the added value of imaging markers in terms of reclassification. Based on a one-year-occurrence rate of subsequent cardiovascular events in the current SMART population database of 2.6%, about 6500 person years of follow-up are needed to obtain the adequate number of endpoints.

ELIGIBILITY:
Inclusion Criteria:

* History of cardiovascular event (coronary carter disease, cardiovascular disease, transient ischemic attack, minor stroke peripheral artery disease , abdominal aortic aneurysm)
* Diabetes Mellitus type 2
* Hypertension (Blood pressure>140/90 mm Hg)

Exclusion Criteria:

* Known renal failure (defined as eGFR <46 ml/min/1.73 m2 estimated based on the modification of diet in renal disease (MDRD) formula)
* Previous allergic reaction to contrast, necessitating medical intervention
* Other contra-indication for CT-scanning (e.g. pregnancy, acute hypotension (<100 mm Hg systolic), clinical instability)
* Prior exposure to ionizing radiation for scientific purposes without advantage for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in consecutive patients entering the SMART study who are eligible according to the in- and exclusion criteria. SMART includes patients aged 18-79 years, who are newly referred to the University Hospital Utrecht with atherosclerotic cardiovascular disease insufficiency will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of cardiovascular events | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
  (non-fatal) ischemic stroke (non-fatal) myocardial infarction (cardio)vascular death Endpoints will be adjudicated by a committee of three experts.

SECONDARY OUTCOMES:
Carotid artery intervention | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
  Carotid desobstruction or stenting
Transient ischemic attack | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
Abdominal aorta aneurysm | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
  Non-fatal rupture, stenting or operation of an abdominal aorta aneurysm
Peripheral artery disease | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
  Amputation, percutaneous transluminal angioplasty or stenting due to peripheral artery disease
Coronary artery intervention | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years
  Percutaneous coronary intervention, coronary artery bypass graft
All cause mortality | Every 26 weeks until death of participant or end of the SMART study, with an expected average of 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda van der Graaf, Prof. dr., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Simons PC, Algra A, van de Laak MF, Grobbee DE, van der Graaf Y. Second manifestations of ARTerial disease (SMART) study: rationale and design. Eur J Epidemiol. 1999 Oct;15(9):773-81. doi: 10.1023/a:1007621514757. PMID 10608355
- [Background] Dorresteijn JA, Visseren FL, Wassink AM, Gondrie MJ, Steyerberg EW, Ridker PM, Cook NR, van der Graaf Y; SMART Study Group. Development and validation of a prediction rule for recurrent vascular events based on a cohort study of patients with arterial disease: the SMART risk score. Heart. 2013 Jun;99(12):866-72. doi: 10.1136/heartjnl-2013-303640. Epub 2013 Apr 10. PMID 23574971